CLINICAL TRIAL: NCT07323108
Title: Investigation of the Effects of Exercises Performed With Stroboscopic Glasses on Athletic Performance in Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KA24/389
Record Dates: First submitted 2025-11-19; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Stroboscopic Glasses
Keywords: volleyball; stroboscopic glasses; physical fitness; sports performance

STUDY DESIGN:
Intervention Model Description: In this study, individuals were evaluated face-to-face at the Beştepe Volleyball Hall of the Turkish Volleyball Federation. Each evaluation lasted 30 minutes. After recording the sociodemographic information of the individuals, they were divided into two groups using a computer numbering system: the stroboscopic glasses group and the control group. The stroboscopic glasses group performed exercises with the glasses. The control group performed exercises without the stroboscopic glasses. The evaluations were conducted three times a week for six weeks, following the players' warm-up exercises. Since only one stroboscopic glasses was used, the evaluations were planned over two days, each lasting 30 minutes. On the first day, reaction time, agility, and anaerobic power were evaluated, respectively; on the second day, coordination and balance were evaluated respectively.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stroboscopic glasses group (Experimental): 20 volleyball players using stroboscopic glasses in training
  Interventions: Device: stroboscopic visual training
- Control group (No Intervention): 20 volleyball players only exercised

INTERVENTIONS:
Device: stroboscopic visual training — 40 volleyball players were evaluated at three times: pre-exercise, after 6 weeks and after 10 weeks regard to reaction time, agility, anaerobic performance, balance and coordination. Experimental group used stroboscopic glasses when doing exercise. Exercise program consisted lunge, jumping and balance exercises. Each exercise consisted 12 repetitions and 3 sets. Stroboscopic glasses were adjusted to 100 ms on/150 ms off flash level 3. This frequency is always preferred scientific research about stroboscopic visual training.
  Arms: stroboscopic glasses group

SUMMARY:
The aim of this study was to examine the effects of exercises performed with stroboscopic glasses on athletic performance in volleyball players. 40 professional male volleyball players aged between 18-35, who had not undergone any surgery in the last 6 months and who had no chronic systemic disease were included in the study. 20 individuals were randomly assigned to the stroboscopic glasses group and 20 individuals to the control group. Individuals in the stroboscopic glasses group were informed about stroboscopic glasses. Individuals in the stroboscopic glasses group wore glasses and individuals in the control group did their exercises without glasses for 6 weeks. Individuals' visual reaction time, auditory reaction time and target-oriented reaction time were measured with the Human Benchmark test, agility assessment with the T Agility test, anaerobic capacity assessment with the vertical jump test, balance assessment with the Flamingo Balance test and coordination assessment with the Hexagonal Coordination test. The evaluations were made three times, before exercise, 6 weeks after exercise and 10 weeks after exercise.

DETAILED DESCRIPTION:
Individuals' visual reaction time, auditory reaction time and target-oriented reaction time were measured with the Human Benchmark test, agility assessment with the T Agility test, anaerobic capacity assessment with the vertical jump test, balance assessment with the Flamingo Balance test and coordination assessment with the Hexagonal Coordination test. The evaluations were made three times, before exercise, 6 weeks after exercise and 10 weeks after exercise.

ELIGIBILITY:
Inclusion Criteria: • Male individuals aged 18-35

* Being a professional volleyball player
* Not having undergone surgery in the last 6 months
* Not having any chronic, systemic, or neuromuscular disease
* Not having visual, cognitive, or vestibular disorders

Exclusion Criteria: • Individuals under 18 and over 35 years of age

* Female individuals
* Sedentary individuals
* Having visual, cognitive, or vestibular disorders

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male volleyball players
Enrollment: 40 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Reaction Time | 10 weeks
  Human Bencmark Test
Agility | 10 weeks
  T Agility Test
Anaerobic performance | 10 weeks
  Vertical Jump Test
Balance | 10 weeks
  Flamingo Balance Test
Coordination | 10 weeks
  Hexagonal Coordination Test

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to privacy policy, volleyball team manager did not want to be shared individual performance data.

REFERENCES:
- [Result] Avedesian JM, Covassin T, Baez S, Nash J, Nagelhout E, Dufek JS. Relationship Between Cognitive Performance and Lower Extremity Biomechanics: Implications for Sports-Related Concussion. Orthop J Sports Med. 2021 Aug 24;9(8):23259671211032246. doi: 10.1177/23259671211032246. eCollection 2021 Aug. PMID 34458386
- [Result] Hulsdunker T, Mierau A. Visual Perception and Visuomotor Reaction Speed Are Independent of the Individual Alpha Frequency. Front Neurosci. 2021 Apr 8;15:620266. doi: 10.3389/fnins.2021.620266. eCollection 2021. PMID 33897344
- [Result] Zwierko T, Tapia V, Vera J, Redondo B, Morenas-Aguilar MD, Garcia-Ramos A. Enhancing reactive agility in soccer: The impact of stroboscopic eyewear during warm-up across fatigued and non-fatigued conditions. Eur J Sport Sci. 2024 Dec;24(12):1798-1808. doi: 10.1002/ejsc.12224. Epub 2024 Nov 22. PMID 39578413
- [Result] Costa E, Gongora M, Bittencourt J, Marinho V, Cagy M, Teixeira S, Nicoliche E, Fernandes I, Machado C, Wienecke J, Ribeiro P, Gupta DS, Velasques B, Budde H. Decrease in reaction time for volleyball athletes during saccadic eye movement task: A preliminary study with evoked potentials. PLoS One. 2024 Jul 3;19(7):e0290142. doi: 10.1371/journal.pone.0290142. eCollection 2024. PMID 38959207